CLINICAL TRIAL: NCT05644223
Title: Effectiveness and Safety of Edaravone Dexborneol in Acute Ischemic Stroke: a Multicenter, Prospective, Patient-centered, Real-world Cohort Study
Brief Title: Effectiveness and Safety of Edaravone Dexborneol in Acute Ischemic Stroke
Acronym: EXPAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Junwei Hao, MD, Director of Neurology Department, Xuanwu Hospital, Beijing
Other Study IDs: SMA-AIS-008
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; edaravone dextrol; real-world study
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposet group: intravenous edaravone dexborneol 37.5mg twice daily
  Interventions: Drug: edaravone dexborneol
- Non-exposed group: standard treatment at the discretion of local clinicians

INTERVENTIONS:
Drug: edaravone dexborneol — intravenous edaravone dexborneol 37.5mg twice daily
  Groups: Exposet group

SUMMARY:
This study is a multicenter, prospective, cohort study to observe the clinical efficacy and safety of edaravone dextrol in patients with acute ischemic stroke in a real-world setting.

DETAILED DESCRIPTION:
The study lasts a total of 90 days and includes three phases: screening, treatment, and follow-up. Treatment period: patients are divided into exposure group and non-exposed group based on the use of edaravone dextrol after ischemic stroke. The exposure group: edaravone dextrol is used according to reference to clinical practice, without specific restrictions. The non-exposed group: edaravone dextrol is not used, and concomitant therapy is at the clinician's discretion. Follow-up period: All patients continue to be followed up to 90 days after stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old；
* Clinically diagnosed as acute ischemic stroke；
* Time from symptom onset to admission≤14 days (symptom onset time is defined as last known well time)；
* Pre-stroke mRS ≤1；
* Have been informed of the content of the informed consent form and agree to participate.

Exclusion Criteria:

* Acute intracranial hemorrhagic diseases confirmed by images: parenchymal hemorrhage, epidural hematoma, subdural hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc.
* Patients who are pregnant or lactating and who are planned to become pregnant within 90 days;
* Patients with severe renal failure (eGFR<30ml/min);
* Patients with concurrent malignancy or severe systemic disease with an estimated survival of less than 90 days;
* Patients with severe mental disorders or unable to complete the informed consent and follow-up due to dementia;
* Patients who are judged unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who aged more than 18 years old and diagnosed as acute ischemic stroke (time from symptom onset to admission ≤ 14 days) with pre-stroke mRS ≤1 can be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 4750 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Scale (mRS) score 0-1 | 90±7 days
  Proportion of patients with modified Rankin Scale (mRS) score (on a scale from 0 to 6, with higher scores indicating greater disability) of 0 to 1 at 90±7 days

SECONDARY OUTCOMES:
Proportion of patients with mRS 0-2 | 90±7 days
  Proportion of patients with mRS score of 0 to 2 at 90±7 days
Distribution of mRS score | 90±7 days
  Distribution of mRS score at 90±7 days
Neurological functional change | at discharge, an average of 7 days
  The change of NIHSS score at discharge compared with the baseline NIHSS score
Quality of Life (EQ-5D-5L) at 90 days | 90±7 days
  The value of EQ-5D-5L at 90±7 days

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage (sICH) | during hospitalization, an average of 7 days
  Symptomatic intracranial hemorrhage during hospitalization
Intracranial hemorrhage during hospitalization (ICH) | during hospitalization
  Intracranial hemorrhage during hospitalization, an average of 7 days
All-cause death | 90±7 days
  All-cause mortality at 90±7 days
Adverse events | during the use of edaravone dexborneol
  Adverse events during the use of edaravone dexborneol

CONTACTS AND LOCATIONS:
Locations (1):
- Junwei Hao, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma G, Raynald, Arham A, Jiang Z, Mo R, Zuo Y, Wu Y, Meng S, Lei S, Nguyen TN, Zhong L; EXPAND investigators. Edaravone Dexborneol in Large Ischemic Stroke: Real-World Experience from a Multicenter Study in China. J Am Heart Assoc. 2026 Jan 6;15(1):e044296. doi: 10.1161/JAHA.125.044296. Epub 2025 Dec 30. PMID 41467380
- [Derived] Ma G, Mo R, Yao X, Nguyen TN, Song Z, Xie W, Yuan G, Zuo Y, Wu Y, Lei S, Meng S, Wu Y, Jiang Z, Liu H, Ren Y, Wang P, Gao D, Chang H, Guo Y, Zhang Q, Ma Q, Zhong L, Song H, Hao J. Clinical and Safety Outcomes of Edaravone Dexborneol in Acute Ischemic Stroke: A Multicenter, Prospective, Cohort Study. Neurology. 2025 Aug 26;105(4):e213949. doi: 10.1212/WNL.0000000000213949. Epub 2025 Aug 5. PMID 40763317